CLINICAL TRIAL: NCT03132532
Title: Phase II Trial of Standard Platinum Doublet Chemotherapy + Various Proton Beam Therapy (PBT) Doses in Order to Determine the Optimal Dose of PBT for Unresectable Stage 2/3 Non-Small Cell Lung Cancer
Brief Title: Platinum Doublet Chemotherapy and Proton Beam Radiation Therapy in Treating Patients With Stage II-III Non-small Cell Lung Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1623; NCI-2017-02481 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16-008343 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2024-01

CONDITIONS: Recurrent Lung Non-Small Cell Carcinoma; Stage II Lung Cancer AJCC v8; Stage III Lung Cancer AJCC v8; Unresectable Lung Non-Small Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Carboplatin; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Etoposide; Paclitaxel; Taxes; Pemetrexed; Proton Therapy; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (platinum doublet chemotherapy, lower dose PBT) (Experimental): Patients receive platinum based doublet chemotherapy consisting of low dose carboplatin and paclitaxel, standard etoposide cisplatin or carboplatin or standard pemetrexed with cisplatin or carboplatin weekly for up to 6 weeks at the discretion of the treating medical oncologist. Patients also undergo lower dose proton beam radiation therapy daily for a total of 60 Gy for up to 30 weekdays in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide; Drug: Paclitaxel; Drug: Pemetrexed; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm C (platinum doublet chemotherapy, higher dose PBT) (Experimental): Patients receive platinum based doublet chemotherapy consisting of low dose carboplatin and paclitaxel, standard etoposide cisplatin or carboplatin or standard pemetrexed with cisplatin or carboplatin weekly for up to 6 weeks at the discretion of the treating medical oncologist. Patients also undergo higher dose proton beam radiation therapy daily for a total of 72 Gy for up to 36 weekdays in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Radiation: Proton Beam Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Carboplatin — Chemotherapy
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cisplatin — Chemotherapy
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm A (platinum doublet chemotherapy, lower dose PBT)
Drug: Etoposide — Chemotherapy
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16; VP 16-213; VP-16; VP-16-213; VP16
  Arms: Arm A (platinum doublet chemotherapy, lower dose PBT)
Drug: Paclitaxel — Chemotherapy
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Pemetrexed — Chemotherapy
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
  Arms: Arm A (platinum doublet chemotherapy, lower dose PBT)
Radiation: Proton Beam Radiation Therapy — Undergo PBT
  Other Names: PBRT; Proton; Proton EBRT; Proton External Beam Radiotherapy; Proton Radiation Therapy; Radiation, Proton Beam
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies how well platinum doublet chemotherapy and proton beam radiation therapy work in treating patients with stage II-III non-small cell lung cancer that cannot be removed by surgery (unresectable). Drugs used in chemotherapy, such as carboplatin, paclitaxel, etoposide, cisplatin, and pemetrexed work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high energy protons to kill tumor cells and shrink tumors. Giving platinum doublet chemotherapy and proton beam radiation therapy may work better in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the 1-year progression-free survival rates of 72 gray (Gy) and 60 Gy conventionally fractionated proton beam therapy (PBT) (as part of concurrent combined modality therapy).

SECONDARY OBJECTIVE:

I. To assess the adverse events, survival, quality of life, and patterns of failure (local regional, distant metastatic) associated with two dose levels of conventionally fractionated PBT (as part of concurrent combined modality therapy).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive platinum based doublet chemotherapy consisting of low dose carboplatin and paclitaxel, standard etoposide cisplatin or carboplatin or standard pemetrexed with cisplatin or carboplatin weekly for up to 6 weeks at the discretion of the treating medical oncologist. Patients also undergo lower dose proton beam radiation therapy daily for a total of 60 Gy for up to 30 weekdays in the absence of disease progression or unacceptable toxicity.

ARM C: Patients receive platinum based doublet chemotherapy consisting of low dose carboplatin and paclitaxel, standard etoposide cisplatin or carboplatin or standard pemetrexed with cisplatin or carboplatin weekly for up to 6 weeks at the discretion of the treating medical oncologist. Patients also undergo higher dose proton beam radiation therapy daily for a total of 72 Gy for up to 36 weekdays in the absence of disease progression or unacceptable toxicity.

All patients undergo computed tomography (CT) throughout the study, magnetic resonance imaging (MRI) or CT, and positron emission tomography (PET)/CT during screening.

After completion of study treatment, patients are followed up every 3 months for 3 years and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Histological confirmation of non-small cell lung cancer
* Forced expiratory volume in 1 second (FEV1) > 1.0 L
* Unresectable or medically inoperable stage 2-3 non-small cell lung cancer (based on computed tomography/positron emission tomography [CT/PET], magnetic resonance imaging [MRI] or CT of brain, and physical exam);

  * Eligible if recurrence after surgery and now has the equivalent stage 2-3 non-small cell lung cancer (NSCLC) OR had sub totally resected stage 2-3 NSCLC
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* White blood cell (WBC) >= 3.0 x 10^9/L
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Hemoglobin (Hgb) >= 9 g/dl
* Platelets (plts) > 100 x 10^9/L
* Serum creatinine < 1.5 x upper limits of normal (ULN)
* Serum bilirubin < 1.5 x ULN
* Provide informed written consent
* Willing to return to enrolling institution for follow-up for a minimum of 1 year
* Ability to undergo potentially curative chemotherapy plus radiotherapy

Exclusion Criteria:

* Any of the following because this study involves an agent that has known genotoxic, mutagenic and teratogenic effects:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Weight loss of > 10% in the past 3 months
* Distant metastases (M1 disease)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, lupus, usual interstitial pneumonitis (UIP), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any investigational agent, that would be considered as a treatment for the primary neoplasm
* Active second malignancy
* History of myocardial infarction =< 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* Received chemotherapy for lung cancer within 6 months of registration
* Previous chest radiotherapy that would overlap with the proton field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2023-12-23 (Actual); Study Completion 2023-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terence T. Sio, M.D., M.S., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT): Patients receive platinum based doublet chemotherapy consisting of low dose carboplatin and paclitaxel, standard etoposide cisplatin or carboplatin or standard pemetrexed with cisplatin or carboplatin weekly for up to 6 weeks at the discretion of the treating medical oncologist. Patients also undergo lower dose proton beam radiation therapy daily for a total of 60 Gy for up to 30 weekdays in the absence of disease progression or unacceptable toxicity.> > Carboplatin: Chemotherapy>
  > Cisplatin: Chemotherapy>
  > Etoposide: Chemotherapy>
  > Paclitaxel: Chemotherapy>
  > Pemetrexed: Chemotherapy>
  > Proton Beam Radiation Therapy: Undergo PBT>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
- Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT): Patients receive platinum based doublet chemotherapy consisting of low dose carboplatin and paclitaxel, standard etoposide cisplatin or carboplatin or standard pemetrexed with cisplatin or carboplatin weekly for up to 6 weeks at the discretion of the treating medical oncologist. Patients also undergo higher dose proton beam radiation therapy daily for a total of 72 Gy for up to 36 weekdays in the absence of disease progression or unacceptable toxicity.>
  > Carboplatin: Chemotherapy>
  > Paclitaxel: Chemotherapy>
  > Proton Beam Radiation Therapy: Undergo PBT>
  > Quality-of-Life Assessment: Ancillary studies>
  > Questionnaire Administration: Ancillary studies
Period: Overall Study
Arm/Group | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT)
Started | 10 | 10
Completed | 10 | 7
Not Completed | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT) | Total
Number analyzed (Participants) | 10 | 7 | 17
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 75.50 [71.50 to 79.50] | 74.0 [69.50 to 78.0] | 74.0 [70.0 to 80.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 7 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Method of Payment [Count of Participants; unit: Participants]
  MEDICARE | 9 | 5 | 14
  MEDICARE AND PRIVATE INSURANCE | 1 | 0 | 1
  PRIVATE INSURANCE | 0 | 2 | 2
Height (Cm) [Mean (Standard Deviation); unit: cm] | 167.100 (11.799) | 171.714 (10.965) | 169.000 (11.352)
Weight (Kg) [Mean (Standard Deviation); unit: Kg] | 73.460 (13.422) | 84.900 (18.190) | 78.171 (16.096)
Smoking Cessation [Count of Participants; unit: Participants]
  Quit | 8 | 5 | 13
  Kept smoking | 2 | 1 | 3
  Non-smoker | 0 | 1 | 1
Baseline QOL [Count of Participants; unit: Participants] — QOL score that can be collected in a minute or so by having each patient judge the overall quality of their lives with a single 0-100 scale. Higher is better.
  Participants
    60 | 0 | 1 | 1
    70 | 0 | 2 | 2
    80 | 2 | 0 | 2
    90 | 5 | 3 | 8
    100 | 3 | 1 | 4
ECOG Performance Status [Count of Participants; unit: Participants] — 0: Fully active, able to carry on all pre-disease performance without restriction
  1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work 0 is better than 1 Population: One patient on Arm C is missing ECOG data
  Participants
    0: number analyzed (Participants) | 10 | 6 | 16
    0 | 3 | 3 | 6
    1: number analyzed (Participants) | 10 | 6 | 16
    1 | 7 | 3 | 10
Mayo prognostic score [Count of Participants; unit: Participants] — The score for each prognostic factor totaled up to a score into a category of of 32-37, 38-43, 44-47, 48-52. Lower is better
  Participants
    32-37 | 0 | 1 | 1
    38-43 | 4 | 3 | 7
    44-47 | 4 | 2 | 6
    48-52 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Progression Free Survival (PFS)
Description: A Cox proportional hazards model stratified by stratification factors will be used to model PFS as a function of dose to test for an overall dose effect (a one-sided p-value < 0.10 will be considered as significant evidence of a dose effect). Subsequently, separate Cox models stratified by stratification factors will compare PFS between 72 Gy and 60 Gy (for each, a one-sided p-value < 0.10 will be considered as significant evidence of superiority). Kaplan Meier estimates and curves by dose level will also be generated
Time Frame: From randomization to the earliest date of documentation of disease progression or death due to any cause, assessed up to 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT): Patients receive platinum based doublet chemotherapy consisting of low dose carboplatin and paclitaxel, standard etoposide cisplatin or carboplatin or standard pemetrexed with cisplatin or carboplatin weekly for up to 6 weeks at the discretion of the treating medical oncologist. Patients also undergo lower dose proton beam radiation therapy daily for a total of 60 Gy for up to 30 weekdays in the absence of disease progression or unacceptable toxicity.
  >
  > Carboplatin: Chemotherapy
  >
  > Cisplatin: Chemotherapy
  >
  > Etoposide: Chemotherapy
  >
  > Paclitaxel: Chemotherapy
  >
  > Pemetrexed: Chemotherapy
  >
  > Proton Beam Radiation Therapy: Undergo PBT
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
- Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT): Patients receive platinum based doublet chemotherapy consisting of low dose carboplatin and paclitaxel, standard etoposide cisplatin or carboplatin or standard pemetrexed with cisplatin or carboplatin weekly for up to 6 weeks at the discretion of the treating medical oncologist. Patients also undergo higher dose proton beam radiation therapy daily for a total of 72 Gy for up to 36 weekdays in the absence of disease progression or unacceptable toxicity.
  >
  > Carboplatin: Chemotherapy
  >
  > Paclitaxel: Chemotherapy
  >
  > Proton Beam Radiation Therapy: Undergo PBT
  >
  > Quality-of-Life Assessment: Ancillary studies
  >
  > Questionnaire Administration: Ancillary studies
Arm/Group | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT)
Number analyzed (Participants) | 10 | 7
proportion of participants | 0.6 [0.362 to 0.995] | 0.429 [0.182 to 1.00]

2. Secondary Outcome: Overall Survival (OS)
Description: Will be modeled using Cox models. Kaplan-Meier estimates and curves by dose level will also be generated. OS will again be analyzed as exploratory analysis after 50 deaths per primary pairwise comparison have occurred or after all patients have completed follow-up (whichever occurs first).
Time Frame: From randomization to death due to any cause, assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT)
Number analyzed (Participants) | 10 | 7
Participants
  Alive | 4 | 2
  Dead | 6 | 5

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Graded by National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Adverse events are graded on a scale of 0-5 with 5 being worst. The number of participants with Grade 2 or higher adverse events will be reported.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT)
Number analyzed (Participants) | 10 | 7
Participants
  AE Grade 2+ | 9 | 6
  AE Grade 3+ | 6 | 5

4. Secondary Outcome: Proportion of Participants With Local-regional Failure
Description: Defined as the proportion of participants with documentation of local recurrence. The cumulative incidence of local failure will be estimated using Gray's methodology and compared across dose levels using Fine-Gray quadratic regression (with death as a competing risk).
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT)
Number analyzed (Participants) | 8 | 7
proportion of participants | 0.2 [0.057 to 0.51] | 0.14 [0.026 to 0.51]

5. Secondary Outcome: Proportion of Participants With Distant Metastasis
Description: Defined as the proportion of participants with documentation of distant metastasis. The cumulative incidence of distant metastasis will be estimated using Gray's methodology and compared across dose levels using Fine-Gray quadratic regression (with death as a competing risk).
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT)
Number analyzed (Participants) | 10 | 7
proportion of participants | 0.1 [0.018 to 0.40] | 0.29 [0.08 to 0.64]

6. Other Pre Specified Outcome: Quality of Life Post Treatment
Description: Measured using the single item Linear Analogue Self-Assessment scale. Descriptive statistics by dose level at each time point will include means, standard deviations, medians, and ranges for each scale. Descriptive graphical techniques will include mean plots by dose over time for each scale. Mixed models will be used to compare each scale across dose levels at each post-baseline time point while adjusting for the baseline value of scale. Will graphically explore patterns of missing data and will employ pattern mixture models for longitudinal analyses. The lowest number measuring worst and higher number measuring best outcome.
Time Frame: Up to 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years
Arm/Group | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT)
All-Cause Mortality (participants affected / at risk) | 6/10 | 5/9
Serious Adverse Events (participants affected / at risk) | 5/10 | 5/9
Other Adverse Events (participants affected / at risk) | 10/10 | 7/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) (N=10) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT) (N=9)
Death NOS (General disorders) | 5 (5) | 5 (5)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Platinum Doublet Chemotherapy, Lower Dose PBT) (N=10) | Arm C (Platinum Doublet Chemotherapy, Higher Dose PBT) (N=9)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (8) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 9 (18) | 4 (4)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 7 (15) | 7 (11)
Nausea (Gastrointestinal disorders) | 4 (5) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 8 (16) | 6 (9)
Pain (General disorders) | 2 (2) | 2 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 6 (6) | 7 (7)
Weight loss (Investigations) | 3 (3) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 5 (7) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (16) | 7 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (18) | 5 (7)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-13): https://cdn.clinicaltrials.gov/large-docs/32/NCT03132532/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT03132532/ICF_001.pdf